CLINICAL TRIAL: NCT02724215
Title: Effect of Sleep Apnea on Blood Pressure Control and Outcome Early After Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Sebastian Zaremba, Physician, University Hospital, Bonn
Other Study IDs: 025/16
Record Dates: First submitted 2016-03-01; First posted 2016-03-31 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Subarachnoid Hemorrhage; Sleep Apnea
Keywords: Subarachnoid hemorrhage; Sleep Apnea
MeSH Terms: conditions — Subarachnoid Hemorrhage; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Sleep Apnea: Patients with increased apnea-hypopnea-index (>5/h)
  Interventions: Device: Sleep Apnea Screening (Out of Center Polysomnography Device)
- Patients without Sleep Apnea: Patients with normal apnea-hypopnea-index (5/h and below)
  Interventions: Device: Sleep Apnea Screening (Out of Center Polysomnography Device)

INTERVENTIONS:
Device: Sleep Apnea Screening (Out of Center Polysomnography Device)

SUMMARY:
In this observational study patients with subarachnoid hemorrhage (SAH) will be screened for sleep apnea (SA) to investigate if SA is associated with impaired blood pressure control and worse clinical outcome early after SAH.

DETAILED DESCRIPTION:
Patients admitted with non-traumatic SAH will be consented and screened for sleep apnea within 48 hours after hospital admission. Blood pressure and clinical outcome will be monitored throughout ICU treatment and hospital stay, respectively. Diagnosis of sleep apnea will be confirmed on follow-up 3-6 month after SAH by sleep apnea screening (portable cardiorespiratory monitoring and out-of-center polysomnography, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid Hemorrhage (Hunt & Hess 1 to 4)
* > 18 years of age
* Ability to consent for study of healthcare proxy able to confirm patient will to participate

Exclusion Criteria:

* Stoke within 3 month prior to admission
* Intubation prior or within 24 hours after admission
* no healthcare proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Subarachnoid Hemorrhage admitted to a University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Time to blood pressure target | Within 10 Days of hospital admission with subarachnoid hemorrhage
  The time required to reach blood pressure target as defined by care provider.
Medication needed to achieve blood pressure target | Within 10 Days of hospital admission with subarachnoid hemorrhage
  Blood pressure medication required to reach blood pressure target as defined by care provider.

SECONDARY OUTCOMES:
Change in modified ranking scale (mRS) from baseline to discharge and follow-up visit, respectively. | 3 to 6 Month after SAH
  Change in modified ranking scale at hospital discharge and at follow-up (3-6 month after SAH) will be assessed and compared between patients with and without sleep apnea. The change from baseline to discharge/follow-up will be compared between groups.
Change in NIH stroke scale score (NIHSS) from admission to discharge and follow-up visit, respectively. | 3 to 6 Month after SAH
  Neurological outcome measured as score in NIHSS at hospital discharge and at follow-up (3-6 month after SAH) will be assessed and compared between patients with and without sleep apnea. The change from baseline to discharge/follow-up will be compared between groups.
Barthel Index at discharge at follow-up visit, respectively. | 3 to 6 Month after SAH
  Impairment of daily living (score in Barthel index) at discharge and at follow-up visit (3 to 6 month after SAH) will be assessed. The change from baseline to discharge/follow-up will be compared between groups.

OTHER OUTCOMES:
Incidence of Sleep Apnea in Patients with Subarachnoid Hemorrhage | 6 Month after SAH

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Gueresir, MD, PhD, Principal Investigator — Vice Chair of Department of Neurosurgery; Sebastian Zaremba, MD, Principal Investigator — Physician
Locations (1):
- Department of Neurology and Department of Neurosurgery, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaremba S, Albus L, Vatter H, Klockgether T, Guresir E. Poor blood pressure control following subarachnoid hemorrhage in patients with sleep apnea. Sleep Breath. 2021 Jun;25(2):777-785. doi: 10.1007/s11325-020-02184-0. Epub 2020 Sep 14. PMID 32926343